CLINICAL TRIAL: NCT04654819
Title: Analysis of Student Confidence Levels and Application Success Rates in Simulator Based Dental Anesthesia Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cahit UCOK, Prof. Dr., Ankara University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AnkaraU 14/16
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Confidence, Self
Keywords: Dental anesthesia; Dental education; Simulators; Technology

STUDY DESIGN:
Who Masked: Participant
Masking Description: The control group did not have access to simulators during the period of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This group made anesthesia application on patients without training on simulators.
- Study group (Experimental): This group made anesthesia application on patients after training on simulators.
  Interventions: Device: Dental anesthesia simulator usage

INTERVENTIONS:
Device: Dental anesthesia simulator usage — Training on dental anesthesia simulator
  Arms: Study group

SUMMARY:
The present study investigates confidence levels reported among intern dentists who used dental anesthesia simulators, before performing local anesthesia on patients as well as patient reports on intern dentist confidence levels to deliver anesthesia injections and compare them to those who did not receive dental anesthesia simulator education. Application success rates will also be investigated and compared.

The study was carried out in the dental anesthesia simulator laboratory and in the faculty clinics of Ankara University, Faculty of Dentistry. A hundred volunteer intern dentists who completed the third year of the 5-year undergraduate education program and who had not performed local anesthesia on a patient contributed. Seventy intern dentists received training on dental anesthesia simulators, and made applications on patients, while 30 intern dentists made applications without training on the dental anesthesia simulators and served as control. With a prepared single questionnaire, intern dentists made self-assessment of preparedness and confidence, educators made assessment of application success rates and treated patients evaluated intern dentists' confidence levels.

DETAILED DESCRIPTION:
Ethical approval was obtained from the Ankara University Faculty of Dentistry Clinical Research Ethics Committee (Approval no: 14/16). The study was carried out in the dental anesthesia simulator laboratory and in the faculty clinics of Ankara University, Faculty of Dentistry within a 2-year period. During the first year of the study, the faculty did not have DAS availability. During this first year 30 intern dentists who had completed the third year of the 5-year undergraduate education program and who could not receive DAS training before their first anesthesia application on a patient, were recruited as a control group among consent to participate. During the second year of the study after DAS became available, 70 intern dentists who had completed the third year of the 5-year undergraduate education program and who had not applied local anesthesia to a patient, were recruited as a study group among consent to participate. The study group applied their first anesthesia application on a patient after DAS education.

For the study 10 conduction anesthesia models mounted on metal rods, (CAM SUG2005-UL-SP, Nissin Dental Products Kyoto, Japan, Figure.1), were provided. The part-task simulators had 11 anesthetic contact sensor points (7 in the upper jaw and 4 in the lower jaw) with 32 anatomically shaped teeth, audio signal and light signal indicators when correct position and angle was achieved. The models had clear pink upper and lower gingivae allowing view of injection, making it ideal for beginner intern dentists, while allowing a more realistic training experience.

Both groups attended theoretical presentations an interactive lesson about IANB from an oral and maxillofacial surgery professor. Technical information about DAS were also covered for the study group lessons. Following lessons, both groups answered a questionnaire concerning preparedness. Afterwards, intern dentists in the control group carried on with patient application whereas the study group carried on with DAS education before continuing on patients.

During DAS lessons the intern dentists applied IANB on simulators. The illumination of the light and sound indicator on the model as a result of injection to the pterygomandibular region was accepted as a successful application. The results of the first five IANB applications made by the intern dentists were recorded. Intern dentists who completed the DAS training completed a questionnaire.

After trainings, both groups applied IANB to a patient for the first time in the clinic and completed another questionnaire. The intraoperative and immediate postoperative complications were monitored. Tingling sensation on the lip and tongue, reported by the patient, was accepted as criteria for profound anesthesia. After achieving anesthesia, the questionnaire, was answered by the patient on whom the application was performed.

Questionnaire:

Section 1: Expectations After Theoretical Education

* The theoretical training adequately prepared me for my first anesthesia application. *
* I feel ready for my first anesthesia application. * Section 2: Expectations After DASM Training
* The DASM training adequately prepared me for my first anesthesia application. *
* I feel ready for my first anesthesia application. *
* It was useful to work on the DASM before my first anesthesia application. * Section 3: IANB application
* Explain if complications developed during anesthesia application.
* I was nervous during anesthesia application. *
* I was sure of myself during anesthesia application. *
* I was confident in determining the front edge of the mandible. *
* I was sure of myself when determining the area to enter the dental injector. *
* I was sure of myself as the dental injector entered soft tissue. *
* I was sure of myself as the dental injector progressed through the soft tissue. *
* I felt that the dental injector touched the mandible. *
* I provided anesthesia. **
* I do not need surveillance in my next application. *
* It was/would have been useful to work on the DASM before my first anesthesia application. * Section 4: To be filled out by your patient
* The intern dentist was confident. *
* The intern dentist gave me confidence. *
* The sting of the needle was painful. *
* The injection of the solution was painful. *
* I felt tingling on my lip. **
* I felt tingling in my tongue. **

  * Questions with answer key: Strongly agree, Agree, Indecisive, Disagree, Strongly disagree.

    * Questions with answer key: Strongly agree, Indecisive, Strongly disagree.

ELIGIBILITY:
Inclusion Criteria:

1. Intern dentists who had completed the third year of the 5-year undergraduate education program
2. Not applied local anesthesia to a patient
3. Consent to participate

Exclusion Criteria:

1. Applied local anesthesia to a patient
2. Not consenting to participate

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Self-reported preparedeness and confidence levels of intern dentists | 2 years
  Intern preparedeness and confidence levels was assesed with a questionnaire answered by the intern dentists. Questions will be answered on a 5 point scale: Strongly agree, Agree, Indecisive, Disagree, Strongly disagree.
Patients perception of intern dentist confidence levels | 2 years
  Patients perception of intern dentist confidence was assesed with a prepared questionnaire answered by the patients. Questions will be answered on a 5 point scale: Strongly agree, Agree, Indecisive, Disagree, Strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Cahit Üçok, Prof. Dr., Study Director — Ankara University
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Turkey (Türkiye)